CLINICAL TRIAL: NCT01810315
Title: Influence of Female Reproductive Cycle and Menopause on Cervicovaginal Tissue Susceptibility to HIV-1 Infections and Tenofovir 1% Gel Activity
Brief Title: Influence of Reproductive Cycle and Menopause on HIV-1 Infection and TFV Gel Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: A12-124
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Baseline (No Intervention): Premenopausal women will undergo baseline sampling in each the follicular and luteal phase. Postmenopausal women will undergo baseline sampling one time.
- TFV 1% Gel (Experimental): Participants will vaginally insert 1 applicator of TFV gel followed by a 2nd applicator 2 hours later. Each applicator contains 4.4 gm of TFV 1% gel.
  Premenopausal women will undergo sampling after TFV gel use in each the follicular and luteal phase. Postmenopausal women will undergo sampling after TFV gel use one time.
  Interventions: Drug: TFV 1% gel
- Estradiol Vaginal Cream (Experimental): Post menopausal women only: Participants will insert 2 grams of estradiol cream into the vagina every night for 14 days and then one gram of estradiol cream into the vagina every other night
  Interventions: Drug: Estradiol vaginal cream
- TFV 1% gel and estradiol cream (Experimental): Postmenopausal women only: Participants will vaginally insert 1 applicator of TFV gel followed by a 2nd applicator 2 hours later. Each applicator contains 4.4 gm of TFV 1% gel. In addition, participants will one gram of estradiol cream into the vagina every other night.
  Interventions: Drug: TFV 1% gel; Drug: Estradiol vaginal cream

INTERVENTIONS:
Drug: TFV 1% gel
  Arms: TFV 1% Gel; TFV 1% gel and estradiol cream
Drug: Estradiol vaginal cream
  Arms: Estradiol Vaginal Cream; TFV 1% gel and estradiol cream

SUMMARY:
Purpose of the study is to assess tenofovir (TFV) PK and PD endpoints, cervicovaginal safety parameters, susceptibility to HIV-1 infection, and objective measures of vaginal applicator use in premenopausal and postmenopausal women.

DETAILED DESCRIPTION:
Premenopausal women: Baseline blood and genital samples will be taken in the follicular and luteal phase (visits 2 and 3). The participant will be given TFV gel and instructed to insert two doses, separated by 2 hours, and return to the clinic 3 hours after the second insertion for blood and genital samples (visits 4/4a and 5/5a).

Postmenopausal women: Premenopausal women: Baseline blood and genital samples will be taken (visit 2). The participant will be given TFV gel and instructed to insert two doses, separated by 2 hours, and return to the clinic 3 hours after the second insertion for blood and genital samples (visit 3/3a). Estradiol cream will be distributed at visit 4. Post estradiol blood and genital samples will be taken at Visit 5. The participant will given TFV gel and instructed to insert 2 doses as before, while continuing to use the estradiol cream. Post TFV gel and estradiol cream blood and genital samples will be taken (visit 6/6a).

ELIGIBILITY:
Inclusion Criteria: All volunteers

* In good healthsignificant systemic disease
* Not at risk of an STI, meaning: In a monogamous heterosexual or same sex relationship for at least the last four months with a partner who is not known to be HIV positive and has no known risks for STIs OR sexually abstinent
* Willing and able to comply with study procedures
* Normal Pap smear (by written report) in the past year.

Inclusion Criteria: Premenopausal volunteers

* 21-to-45 years of age
* Not at risk for pregnancy, meaning:
* Regular menstrual cycles (every 24 - 35 days)
* Luteal phase P level of greater than or equal to 3 ng/ml

Inclusion Criteria: Postmenopausal volunteers

* 46-89 years of age OR both ovaries removed at least 30 days prior to Visit 1
* No menstrual periods/vaginal bleeding in the past 12 months OR both ovaries removed at least 30 days prior to Visit 1
* FSH level of greater than or equal to 20 MIU/ml

Exclusion Criteria: All volunteers

* Clinically significant history of an abnormal Pap smear in the past year
* Surgery or biopsy of the vagina or cervix within 30 days
* Current STI or lower genital tract infection
* Current use of chronic immunosuppressants
* Current presence of vulvar, anal and/or vaginal genital warts
* Current tobacco use of any amount
* History of sensitivity/allergy to any component of the study product, topical anesthetic, or allergy to silver nitrate and/or Monsel's solution
* Known bleeding disorder that could lead to prolonged or continuous bleeding
* Grade 1 or higher laboratory abnormality, per the August 2009 update of the DAIDS Table for Grading the Severity of Adverse Events
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals, antivirals or antiretrovirals.
* Investigator discretion
* Current participation in any other drug or device study

Exclusion Criteria: Premenopausal women

* Use of DMPA in last six months
* Use of any other hormonal contraceptive method without 2 subsequent, normal menses since stopping hormonal contraceptives
* Current use of copper IUD
* Currently pregnant or pregnancy within the past 3 months
* Currently breastfeeding/having breastfed an infant in the last 2 months

Exclusion Criteria: Postmenopausal women

* Use of any hormonal medications in the past 30 days
* Contraindications to vaginal estrogen cream

Ages: 21 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Concentrations of tenofovir in plasma, vaginal aspirate, and genital tissue | 3 hours after dosing
Concentrations of TFV-DP in genital tissue | 3 hours after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Eastern Virginia Medical School, Norfolk, Virginia, United States